CLINICAL TRIAL: NCT00127400
Title: A Pilot Study Comparing the Efficacy of Group Versus Individual Anger Management in Subjects With Intermittent Explosive Disorder
Brief Title: A Pilot Study Comparing the Efficacy of Group Versus Individual Anger Management in Subjects With IED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 11487A
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Anger; Intermittent Explosive Disorder
Keywords: anger; intermittent; explosive
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders | interventions — Anger Management Therapy

INTERVENTIONS:
Behavioral: anger management therapy

SUMMARY:
The purpose of this study is to see how different forms of "Anger Management" compare in reducing anger and impulsive aggressive symptoms in people. "Anger Management" is a common form of "talk therapy" used to help people with anger problems. There are different types of "talk therapy" used to help people for anger problems and this study will compare two types of talk therapy in people with Intermittent Explosive Disorder (IED). IED is a disorder in which there are frequent and sudden outbursts of anger (yelling, throwing and breaking things, hitting people) that lead to problems with other people socially or at work.

DETAILED DESCRIPTION:
Intermittent Explosive Disorder (IED) is increasingly acknowledged as a common, potentially disabling psychiatric condition. Despite this, there are currently no empirically supported behavioral treatments for patients with IED. The purpose of the proposed study is to assess the short-term and long-term efficacy of a cognitive-behavioral treatment (CBT), previously found to be successful in treating dysfunctional anger, for treating IED. Secondary goals of the project are to:

1. explore mechanisms involved in the successful treatment of IED, and
2. examine individual differences associated with treatment response.

Seventy-two subjects meeting for both research and DSM IED criteria will be randomly assigned to either 12 weeks of individual CBT, 12 weeks of group CBT or 12 weeks of a wait-list control condition. Subjects will be assessed before and after therapy/wait-list as well as at 3 month and 6 month follow-up. Primary outcome measures will assess aggressive behavior, anger, and the presence of an IED diagnosis at post-treatment, 6-month follow-up and 12-month follow-up. Social and emotional information processing will be evaluated as potential mechanism of change. Trait aggression will be assessed as a potential moderating variable.

ELIGIBILITY:
Inclusion Criteria:

* The subject meets research criteria for a lifetime diagnosis of intermittent explosive disorder (IED).
* The subject has a Trait Anger Score > 21 on the STAXI (see above).
* Subject is willing to be randomized to any one of the four conditions.
* The subject is willing and able to cooperate with study protocol (i.e., keep appointments, complete rating forms, etc.)
* Subject gives informed consent to participate in study.

Exclusion Criteria:

* The subject has any history of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) Axis I bipolar mood disorder, schizophrenia, delusional disorder, organic brain disorder, mental retardation.
* The subject meets DSM-IV criteria for alcohol or drug dependence within 30 days prior to the start of any of the study conditions.
* The subject has a Beck Depression Inventory, 2nd Edition (BDI-II) score > 32.
* The subject has aggressive obsessions in the context of Obsessive Compulsive Disorder (OCD).
* Current suicidal behavior or homicidal ideation.
* The subject is not willing to be randomized to any one of the four conditions.
* The subject is not willing to cooperate with study protocol (i.e., keep appointments, complete rating forms, etc.).
* The subject, in the opinion of the principal investigator (PI), is not able or likely to cooperate with study protocol (i.e., keep appointments, complete rating forms, etc.)
* The subject is already engaged in an anger management program elsewhere.
* The subject does not give informed consent to participate in study

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72
Dates: Start 2002-02; Study Completion 2006-07

PRIMARY OUTCOMES:
Aggression interview (Overt Aggression Scale-Modified
[OASM]) at midpoint 1 week post-treatment, 3-month follow-up and 6-month follow-up
State-Trait Anxiety Inventory (STAXI) questionnaire at midpoint 1 week post-treatment, 3-month follow-up and 6-month follow-up

SECONDARY OUTCOMES:
Behavioral aggression measures (Taylor Aggression Paradigm [TAP], Point Subtraction Aggression Paradigm [PSAP]) at 1 week post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael McCloskey, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Deffenbacher JL, Filetti LB, Lynch RS, Dahlen ER, Oetting ER. Cognitive-behavioral treatment of high anger drivers. Behav Res Ther. 2002 Aug;40(8):895-910. doi: 10.1016/s0005-7967(01)00067-5. PMID 12186353
- [Background] Deffenbacher, J. L., & McKay, M. (2000). Overcoming Situational and General Anger: A protocol for the treatment of anger based on relaxation, cognitive restructuring, and coping skills training. New Harbinger Publication: Oakland
- [Background] Deffenbacher, J. L., McNamara, K., Stark, R. S., & Sabadell, P. M. (1990a). A comparison of cognitive-behavioral and process-oriented group counseling for general anger reduction. Journal of Counseling & Development, 69, 167-69.
- [Background] Deffenbacher, J. L., McNamara, K., Stark, R. S., & Sabadell, P. M. (1990b). A combination of cognitive, relaxation, and behavioral coping skills in the reduction of general anger. Journal of College Student Development, 31, 351-358.
- [Background] Deffenbacher, J. L., Oetting, E. R., Huff, M. E., Cornell, G. R., & Dallager, C. J. (1996a). Evaluation of two cognitive-behavioral approaches to general anger reduction. Cognitive Therapy and Research, 20, 551-573.
- [Background] Deffenbacher, J. L., Oetting, E. R., Huff, M. E., & Thwaites, G. A. (1995). Fifteen-month follow-up of social skills and cognitive-relaxation approaches to general anger reduction. Journal of Counseling Psychology, 42, 400-405.
- [Background] Deffenbacher JL, Oetting ER, Lynch RS, Morris CD. The expression of anger and its consequences. Behav Res Ther. 1996 Jul;34(7):575-90. doi: 10.1016/0005-7967(96)00018-6. PMID 8826765
- [Background] Deffenbacher, J. L., & Stark, R. S. (1992). Relaxation and cognitive-relaxation treatments of general anger. Journal of Counseling Psychology, 39, 158-167.
- [Background] DiGiuseppe, R. & Tafrate, R. C. (2003). Anger Treatment for Adults: A Meta-Analytic Review. Clinical Psychology Science & Practice, 10, 70-84.